CLINICAL TRIAL: NCT00980200
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Five Period Cross-over Study to Evaluate the Efficacy and Safety of Selected Doses and Dose Intervals of GW642444 Administered Via a Novel Dry Powder Inhaler (NDPI) in Subjects ≥18 Years of Age With Persistent Asthma
Brief Title: Efficacy and Safety Study in Subjects With Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 113310
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Results first posted 2013-08-07 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2016-12

CONDITIONS: Asthma
Keywords: GW642444; once daily dosing; asthma; efficacy; safety; FEV1
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- C/E/A/B/D (Experimental): GW642444 Dose 2 QD/GW642444 Dose 4 QD/placebo/GW642444 Dose 1 BD/GW642444 Dose 3 QD
  Interventions: Drug: Dose 2 QD
- D/C/E/A/B (Experimental): GW642444 Dose 3 QD/GW642444 Dose 2 QD/GW642444 Dose 4 QD/placebo/GW642444 Dose 1 BD
  Interventions: Drug: Dose 3 QD
- A/B/C/D/E (Experimental): placebo/GW642444 Dose 1 BD/GW642444 Dose 2 QD/GW642444 Dose 3 QD/GW642444 Dose 4 QD
  Interventions: Drug: placebo
- B/A/D/E/C (Experimental): GW642444 Dose 1 BD/placebo/GW642444 Dose 3 QD/GW642444 Dose 4 QD/GW642444 Dose 2 QD
  Interventions: Drug: Dose 1 BD
- E/D/B/C/A (Experimental): GW642444 Dose 4 QD/GW642444 Dose 3 QD/GW642444 Dose 1 BD/GW642444 Dose 2 QD/placebo
  Interventions: Drug: Dose 4 QD

INTERVENTIONS:
Drug: Dose 4 QD — QD once daily
  Arms: E/D/B/C/A
Drug: Dose 3 QD — QD once daily
  Arms: D/C/E/A/B
Drug: placebo — placebo
  Arms: A/B/C/D/E
Drug: Dose 2 QD — QD once daily
  Arms: C/E/A/B/D
Drug: Dose 1 BD — BD twice daily
  Arms: B/A/D/E/C

SUMMARY:
The study is a multi-center, double-blind, placebo-controlled, cross-over study to evaluate the efficacy and safety of selected doses and dose intervals of the novel long acting beta agonist (LABA), GW642444 in asthmatic subjects ≥18 years of age who are currently receiving inhaled corticosteroid treatment.

DETAILED DESCRIPTION:
The study will be a five-period cross-over study with each 7 day treatment period separated by a 7 day wash-out period. The study will enroll asthmatic subjects ≥18 years of age who are currently receiving inhaled corticosteroid treatment with an FEV1 of between 40-85% of predicted normal and with airway reversibility as demonstrated by an increase in FEV1 of ≥12% and ≥200ml .

Efficacy assessments include 24-hour serial lung function testing. Safety assessments include incidence of adverse events and measurement of vital signs.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient
* ≥18 years of age at Visit 1
* Male or Eligible Female
* Diagnosis of asthma at least 12 weeks prior to Visit 1
* Disease reversibility
* Current anti-asthma therapy
* Appropriately signed and dated informed consent has been obtained
* Able to comply with all the study requirements

Exclusion Criteria:

* History of Life-Threatening Asthma
* No use of systemic corticosteroids for any indication within 8 weeks prior to Visit
* No concurrent diseases/abnormalities that would put the safety of the subject at risk through study participation
* Drug Allergy to β2 agonist or sympathomimetic drugs, or known or suspected sensitivity to lactose or magnesium stearate
* History of severe milk protein allergy
* Non-compliance with study medication and other study-related requirements
* No use of inhaled tobacco products within the past three months or historical use of 10 pack years or more
* Administration of prohibited medications and non-drug therapies and corresponding timeframes as outlined in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2009-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (9):
- United States (9):
  - GSK Investigational Site, Cypress, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Bethesda, Maryland
  - GSK Investigational Site, Rolla, Missouri
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Boerne, Texas

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Sterling R, Lim J, Frith L, Snowise NG, Jacques L, Haumann B. Efficacy and optimal dosing interval of the long-acting beta(2) agonist, vilanterol, in persistent asthma: a randomised trial. Respir Med. 2012 Aug;106(8):1110-5. doi: 10.1016/j.rmed.2012.03.007. Epub 2012 Apr 19. PMID 22520084
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 113310 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113310 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113310 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113310 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113310 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113310 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113310 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (par,) who met all inclusion criteria at screening entered a 7-day Run-in Period (RIP). Par. were instructed to administer albuterol inhalation aerosol as needed and to continue their inhaled corticosteroid at a stable dose throughout the study. Par. who met randomization criteria at the end of the RIP entered Treatment Period 1.
Pre-assignment Details: The study was a multi-centre, double-blind, placebo-controlled, five-period cross-over study. Following the 7(+7)-day RIP, eligible participants were randomized to 1 of 5 sequences of GW642444 at doses of 6.25 micrograms (µg) once daily (QD), 6.25 µg twice daily, 12.5 µg QD, 25 µg QD, and placebo.
Groups:
- Sequence 1: 6.25 µg BID, Pbo, 12.5 µg QD, 25 µg QD, 6.25 µg QD: Participants received GW642444 6.25 micrograms (µg) twice a day (BID), placebo (pbo), GW642444 12.5 µg once a day (QD) in the evening, GW642444 25 µg QD in the evening, and GW642444 6.25 µg QD in the evening in Treatment Periods 1, 2, 3, 4, and 5 respectively. Participants received all treatments from a Dry Powder Inhaler (DPI) for 7 days. The treatments were administered approximately 12 hours apart. All participants took blinded treatment (active or placebo) every 12 hours, and therefore followed a 12-hour dosing interval. The five treatment periods were separated by a washout period of at least 7 days.
- Sequence 2: Pbo, 6.25 µg BID, 6.25 µg QD, 12.5 µg QD, 25 µg QD: Participants received placebo, GW642444 6.25 µg BID, GW642444 6.25 µg QD in the evening, GW642444 12.5 µg QD in the evening, and GW642444 25 µg QD in the evening and in Treatment Periods 1, 2, 3, 4, and 5 respectively. Participants received all treatments from a DPI for 7 days. The treatments were administered approximately 12 hours apart. All participants took blinded treatment (active or placebo) every 12 hours, and therefore followed a 12-hour dosing interval. The five treatment periods were separated by a washout period of at least 7 days.
- Sequence 3: 6.25 µg QD, 25 µg QD, Pbo, 6.25 µg BID, 12.5 µg QD: Participants received GW642444 6.25 µg QD in the evening, GW642444 25 µg QD in the evening, placebo, GW642444 6.25 µg BID, and GW642444 12.5 µg QD in the evening in Treatment Periods 1, 2, 3, 4, and 5 respectively. Participants received all treatments from a DPI for 7 days. The treatments were administered approximately 12 hours apart. All participants took blinded treatment (active or placebo) every 12 hours, and therefore followed a 12-hour dosing interval. The five treatment periods were separated by a washout period of at least 7 days.
- Sequence 4: 12.5 µg QD, 6.25 µg QD, 25 µg QD, Pbo, 6.25 µg BID: Participants received GW642444 12.5 µg QD in the evening, GW642444 6.25 µg QD in the evening, GW642444 25 µg QD in the evening, placebo, and GW642444 6.25 µg BID and in Treatment Periods 1, 2, 3, 4, and 5 respectively. Participants received all treatments from a DPI for 7 days. The treatments were administered approximately 12 hours apart. All participants took blinded treatment (active or placebo) every 12 hours, and therefore followed a 12-hour dosing interval. The five treatment periods were separated by a washout period of at least 7 days.
- Sequence 5: 25 µg QD, 12.5 µg QD, 6.25 µg BID, 6.25 µg QD, Pbo: Participants received GW642444 25 µg QD in the evening, GW642444 12.5 µg QD in the evening, GW642444 6.25 µg BID, GW642444 6.25 µg QD in the evening, and placebo in Treatment Periods 1, 2, 3, 4, and 5 respectively. Participants received all treatments from a DPI for 7 days. The treatments were administered approximately 12 hours apart. All participants took blinded treatment (active or placebo) every 12 hours, and therefore followed a 12-hour dosing interval. The five treatment periods were separated by a washout period of at least 7 days.
Period: 7-day Treatment Period 1
Arm/Group | Sequence 1: 6.25 µg BID, Pbo, 12.5 µg QD, 25 µg QD, 6.25 µg QD | Sequence 2: Pbo, 6.25 µg BID, 6.25 µg QD, 12.5 µg QD, 25 µg QD | Sequence 3: 6.25 µg QD, 25 µg QD, Pbo, 6.25 µg BID, 12.5 µg QD | Sequence 4: 12.5 µg QD, 6.25 µg QD, 25 µg QD, Pbo, 6.25 µg BID | Sequence 5: 25 µg QD, 12.5 µg QD, 6.25 µg BID, 6.25 µg QD, Pbo
Started | 15 | 14 | 15 | 16 | 15
Completed | 15 | 13 | 15 | 16 | 15
Not Completed | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0
Period: 7-day Washout Period 1
Arm/Group | Sequence 1: 6.25 µg BID, Pbo, 12.5 µg QD, 25 µg QD, 6.25 µg QD | Sequence 2: Pbo, 6.25 µg BID, 6.25 µg QD, 12.5 µg QD, 25 µg QD | Sequence 3: 6.25 µg QD, 25 µg QD, Pbo, 6.25 µg BID, 12.5 µg QD | Sequence 4: 12.5 µg QD, 6.25 µg QD, 25 µg QD, Pbo, 6.25 µg BID | Sequence 5: 25 µg QD, 12.5 µg QD, 6.25 µg BID, 6.25 µg QD, Pbo
Started | 15 | 13 | 15 | 16 | 15
Completed | 15 | 13 | 15 | 16 | 15
Not Completed | 0 | 0 | 0 | 0 | 0
Period: 7-day Treatment Period 2
Arm/Group | Sequence 1: 6.25 µg BID, Pbo, 12.5 µg QD, 25 µg QD, 6.25 µg QD | Sequence 2: Pbo, 6.25 µg BID, 6.25 µg QD, 12.5 µg QD, 25 µg QD | Sequence 3: 6.25 µg QD, 25 µg QD, Pbo, 6.25 µg BID, 12.5 µg QD | Sequence 4: 12.5 µg QD, 6.25 µg QD, 25 µg QD, Pbo, 6.25 µg BID | Sequence 5: 25 µg QD, 12.5 µg QD, 6.25 µg BID, 6.25 µg QD, Pbo
Started | 15 | 13 | 15 | 16 | 15
Completed | 15 | 13 | 15 | 16 | 15
Not Completed | 0 | 0 | 0 | 0 | 0
Period: 7-day Washout Period 2
Arm/Group | Sequence 1: 6.25 µg BID, Pbo, 12.5 µg QD, 25 µg QD, 6.25 µg QD | Sequence 2: Pbo, 6.25 µg BID, 6.25 µg QD, 12.5 µg QD, 25 µg QD | Sequence 3: 6.25 µg QD, 25 µg QD, Pbo, 6.25 µg BID, 12.5 µg QD | Sequence 4: 12.5 µg QD, 6.25 µg QD, 25 µg QD, Pbo, 6.25 µg BID | Sequence 5: 25 µg QD, 12.5 µg QD, 6.25 µg BID, 6.25 µg QD, Pbo
Started | 15 | 13 | 15 | 16 | 15
Completed | 15 | 13 | 15 | 16 | 15
Not Completed | 0 | 0 | 0 | 0 | 0
Period: 7-day Treatment Period 3
Arm/Group | Sequence 1: 6.25 µg BID, Pbo, 12.5 µg QD, 25 µg QD, 6.25 µg QD | Sequence 2: Pbo, 6.25 µg BID, 6.25 µg QD, 12.5 µg QD, 25 µg QD | Sequence 3: 6.25 µg QD, 25 µg QD, Pbo, 6.25 µg BID, 12.5 µg QD | Sequence 4: 12.5 µg QD, 6.25 µg QD, 25 µg QD, Pbo, 6.25 µg BID | Sequence 5: 25 µg QD, 12.5 µg QD, 6.25 µg BID, 6.25 µg QD, Pbo
Started | 15 | 13 | 15 | 16 | 15
Completed | 15 | 12 | 15 | 16 | 14
Not Completed | 0 | 1 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0 | 1
Period: 7-day Washout Period 3
Arm/Group | Sequence 1: 6.25 µg BID, Pbo, 12.5 µg QD, 25 µg QD, 6.25 µg QD | Sequence 2: Pbo, 6.25 µg BID, 6.25 µg QD, 12.5 µg QD, 25 µg QD | Sequence 3: 6.25 µg QD, 25 µg QD, Pbo, 6.25 µg BID, 12.5 µg QD | Sequence 4: 12.5 µg QD, 6.25 µg QD, 25 µg QD, Pbo, 6.25 µg BID | Sequence 5: 25 µg QD, 12.5 µg QD, 6.25 µg BID, 6.25 µg QD, Pbo
Started | 15 | 12 | 15 | 16 | 14
Completed | 15 | 12 | 15 | 16 | 14
Not Completed | 0 | 0 | 0 | 0 | 0
Period: 7-day Treatment Period 4
Arm/Group | Sequence 1: 6.25 µg BID, Pbo, 12.5 µg QD, 25 µg QD, 6.25 µg QD | Sequence 2: Pbo, 6.25 µg BID, 6.25 µg QD, 12.5 µg QD, 25 µg QD | Sequence 3: 6.25 µg QD, 25 µg QD, Pbo, 6.25 µg BID, 12.5 µg QD | Sequence 4: 12.5 µg QD, 6.25 µg QD, 25 µg QD, Pbo, 6.25 µg BID | Sequence 5: 25 µg QD, 12.5 µg QD, 6.25 µg BID, 6.25 µg QD, Pbo
Started | 15 | 12 | 15 | 16 | 14
Completed | 15 | 12 | 15 | 16 | 14
Not Completed | 0 | 0 | 0 | 0 | 0
Period: 7-day Washout Period 4
Arm/Group | Sequence 1: 6.25 µg BID, Pbo, 12.5 µg QD, 25 µg QD, 6.25 µg QD | Sequence 2: Pbo, 6.25 µg BID, 6.25 µg QD, 12.5 µg QD, 25 µg QD | Sequence 3: 6.25 µg QD, 25 µg QD, Pbo, 6.25 µg BID, 12.5 µg QD | Sequence 4: 12.5 µg QD, 6.25 µg QD, 25 µg QD, Pbo, 6.25 µg BID | Sequence 5: 25 µg QD, 12.5 µg QD, 6.25 µg BID, 6.25 µg QD, Pbo
Started | 15 | 12 | 15 | 16 | 14
Completed | 15 | 12 | 15 | 16 | 14
Not Completed | 0 | 0 | 0 | 0 | 0
Period: 7-day Treatment Period 5
Arm/Group | Sequence 1: 6.25 µg BID, Pbo, 12.5 µg QD, 25 µg QD, 6.25 µg QD | Sequence 2: Pbo, 6.25 µg BID, 6.25 µg QD, 12.5 µg QD, 25 µg QD | Sequence 3: 6.25 µg QD, 25 µg QD, Pbo, 6.25 µg BID, 12.5 µg QD | Sequence 4: 12.5 µg QD, 6.25 µg QD, 25 µg QD, Pbo, 6.25 µg BID | Sequence 5: 25 µg QD, 12.5 µg QD, 6.25 µg BID, 6.25 µg QD, Pbo
Started | 15 | 12 | 15 | 16 | 14
Completed | 15 | 12 | 15 | 16 | 14
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- PB, GW642444 6.25 µg QD, 6.25 µg BID, 12.5 µg QD, and 25 µg QD: All participants received one of the following five treatments in one of the five Treatment Periods from two DPI dispensed on Day 1of each of the five 7-day treatment periods: Placebo (PB), GW642444 6.25 µg once daily (QD) in the evening, GW642444 6.25 µg twice daily (BID), GW642444 12.5 µg QD in the evening, and GW642444 25 µg QD in the evening. Participants received their first evening medication dose in the clinic on Day 1 of each of the five treatment periods. The treatments were administered in the morning (AM) and in the evening (PM), approximately 12 hours apart. All participants took blinded treatment (active or placebo) every 12 hours, and therefore followed a 12-hour dosing interval. The five treatment periods were separated by a 7-day washout period.
Arm/Group | PB, GW642444 6.25 µg QD, 6.25 µg BID, 12.5 µg QD, and 25 µg QD
Number analyzed (Participants) | 75
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.9 (14.37)
Gender [Count of Participants; unit: Participants]
  Female | 47
  Male | 28
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage | 23
  Asian-Central/South Asian Heritage | 1
  White - White/Caucasian/European Heritage | 51

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough (Pre-bronchodilator and Pre-dose) FEV1 on Day 7 of the Treatment Period
Description: Pulmonary function was measured by forced expiratory volume in one second (FEV1), defined as the maximal amount of air that can be forcefully exhaled in one second. Trough FEV1 is defined as the mean of the FEV1 values obtained at the last two scheduled time points at the Day 7 clinic visit (i.e., 11 and 12 hours after the morning dose, or 23 and 24 hours after the evening dose). Change from Baseline was calculated as the Day 7 value minus the Baseline value. Analysis was performed using a mixed model analysis of covariance (ANCOVA) with fixed effects of treatment, period, sex, and age. Participants is fitted as a random effect, and the period Baseline measurement is included as part of a bivariate response. The model for the period Baseline value is not affected by treatment group.
Time Frame: Baseline and Day 7 of the treatment period (up to Study Day 63)
Population: Intent-to Treat (ITT) Population: all participants randomized to treatment who received at least one dose of trial medication. Randomized participants were assumed to have received trial medication unless definitive evidence to the contrary existed. Only participants available at the indicated time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- Placebo: Participants received 2 placebo actuations per day during one of the five 7-day Treatment Periods. Participants received treatment in the morning (AM) and evening (PM), approximately 12 hours apart, from two seperate DPIs starting with their first dose on the evening of Day 1. Each treatment period was followed by a 7-day washout period.
- GW642444 6.25 µg QD: Participants received 2 actuations per day (AM and PM) during one of the five 7-day Treatment Periods from two seperate DPIs starting with their first dose on the evening of Day 1. Participants received one actuation of GW642444 6.25 µg and another actuation of placebo. The treatments were administered approximately 12 hours apart. All participants took blinded treatment (active or placebo) every 12 hours, and therefore followed a 12-hour dosing interval. Each treatment period was followed by a 7-day washout period.
- GW642444 6.25 µg BID: Participants received 2 actuations per day for during one of the five 7-day Treatment Periods from two separate DPIs starting with their first dose on the evening of Day 1. Participants received one actuation of GW642444 6.25 µg in the morning and a second actuation in the evening. The treatments were administered approximately 12 hours apart. All participants took blinded treatment every 12 hours, and therefore followed a 12-hour dosing interval. Each treatment period was followed by a 7-day washout period.
- GW642444 12.5 µg QD: Participants received 2 actuations per day (AM and PM) during one of the five 7-day Treatment Periods from two seperate DPIs starting with their first dose on the evening of Day 1. Participants received one actuation of GW642444 12.5 µg and another actuation of placebo. The treatments were administered approximately 12 hours apart. All participants took blinded treatment (active or placebo) every 12 hours, and therefore followed a 12-hour dosing interval. Each treatment period was followed by a 7-day washout period.
- GW642444 25 µg QD: Participants received 2 actuations per day (AM and PM) during one of the five 7-day Treatment Periods from two seperate DPIs starting with their first dose on the evening of Day 1. Participants received one actuation of GW642444 25 µg and another actuation of placebo. The treatments were administered approximately 12 hours apart. All participants took blinded treatment (active or placebo) every 12 hours, and therefore followed a 12-hour dosing interval. Each treatment period was followed by a 7-day washout period.
Arm/Group | Placebo | GW642444 6.25 µg QD | GW642444 6.25 µg BID | GW642444 12.5 µg QD | GW642444 25 µg QD
Number analyzed (Participants) | 74 | 73 | 74 | 73 | 73
Liters | 0.059 (0.0221) | 0.153 (0.0222) | 0.198 (0.0221) | 0.161 (0.0221) | 0.184 (0.0221)
Statistical Analysis 1: Comparison: Placebo vs GW642444 6.25 µg QD; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.094, 95% CI 2-sided [0.049 to 0.140]
Statistical Analysis 2: Comparison: Placebo vs GW642444 6.25 µg BID; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.140, 95% CI 2-sided [0.095 to 0.185]
Statistical Analysis 3: Comparison: Placebo vs GW642444 12.5 µg QD; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.102, 95% CI 2-sided [0.057 to 0.147]
Statistical Analysis 4: Comparison: Placebo vs GW642444 25 µg QD; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.125, 95% CI 2-sided [0.080 to 0.170]

2. Secondary Outcome: Change From Baseline in Weighted Mean 24-hour FEV1 on Day 7 of the Treatment Period
Description: Pulmonary function was measured by FEV1, defined as the maximal amount of air that can be forcefully exhaled in one second. Weighted mean was derived by calculating the average area under curve, and then dividing by the relevant time interval. 24-hour serial measurements of FEV1 were performed on Day 7 of each of the 5 treatment periods (Visits 3, 5, 7, 9, and 11). Measurements were taken at pre-dose; 30 and 60 minutes; and 3, 5, 11, 12, 12.5, 13, 15, 17, 23, and 24 hours post-dose. Visits 3, 5, 7, 9, and 11 were overnight visits. Change from Baseline was calculated as the Day 7 value minus the Baseline value. Analysis was performed using a mixed effects analysis of covariance (ANCOVA) model, with fixed effects for treatment, period, sex, and age. Participant was fitted as a random effect, and the period Baseline FEV1 measurement was included as part of a bivariate response. The model for the period Baseline value is not affected by treatment group.
Time Frame: Baseline and Day 7 of the treatment period (up to Study Day 63)
Population: ITT Population. Only those participants available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | GW642444 6.25 µg QD | GW642444 6.25 µg BID | GW642444 12.5 µg QD | GW642444 25 µg QD
Number analyzed (Participants) | 74 | 73 | 74 | 73 | 73
Liters | 0.028 (0.0195) | 0.181 (0.0195) | 0.194 (0.0195) | 0.196 (0.0195) | 0.213 (0.0195)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from randomization until follow-up (up to Day 70).
Description: SAEs and non-serious AEs were reported for members of the Intent-to-Treat (ITT) Population, comprised of all participants randomized to treatment who received at least one dose of trial medication. Randomized participants were assumed to have received trial medication unless definitive
Arm/Group | Placebo | GW642444 6.25 µg QD | GW642444 6.25 µg BID | GW642444 12.5 µg QD | GW642444 25 µg QD
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/73 | 0/74 | 0/73 | 0/73
Other Adverse Events (participants affected / at risk) | 1/74 | 0/73 | 3/74 | 0/73 | 3/73
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=74) | GW642444 6.25 µg QD (N=73) | GW642444 6.25 µg BID (N=74) | GW642444 12.5 µg QD (N=73) | GW642444 25 µg QD (N=73)
Upper respiratory tract information (Infections and infestations) | 1 | 0 | 3 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.